CLINICAL TRIAL: NCT06192615
Title: Minimizing ICU Neurological Dysfunction With Dexmedetomidine-induced Sleep (MINDDS II)
Acronym: MINDDS II
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Anesthetist-in-Chief, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2023P003359
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-01

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Intravenous Dexmedetomidine (Experimental): After admission to the ICU and discontinuation of mechanical ventilation, intravenous dexmedetomidine (1 μg/kg over 40 minutes, a maximal dose of 80 μg) and a sublingual placebo (inert film) will be administered nightly for the first three nights while the patient is in the intensive care unit.
  Interventions: Drug: Intravenous Dexmedetomidine; Drug: Sublingual Placebo
- Sublingual Dexmedetomidine (Experimental): After admission to the ICU and discontinuation of mechanical ventilation, sublingual dexmedetomidine (120 μg) and an intravenous placebo (0.9% saline over 40 minutes) will be administered nightly for the first three nights while the patient is in the intensive care unit.
  Interventions: Drug: Sublingual Dexmedetomidine; Drug: Intravenous Placebo
- Placebo (Placebo Comparator): After admission to the ICU and discontinuation of mechanical ventilation, an intravenous placebo (0.9% saline over 40 minutes) and a sublingual placebo (inert film) will be administered nightly for the first three nights while the patient is in the intensive care unit.
  Interventions: Drug: Intravenous Placebo; Drug: Sublingual Placebo

INTERVENTIONS:
Drug: Intravenous Dexmedetomidine — Intravenous dexmedetomidine (1 μg/kg over 40 minutes, a maximal dose of 80 μg)
  Other Names: Intravenous Precedex
  Arms: Intravenous Dexmedetomidine
Drug: Sublingual Dexmedetomidine — Sublingual dexmedetomidine (120 μg)
  Other Names: Sublingual Precedex
  Arms: Sublingual Dexmedetomidine
Drug: Intravenous Placebo — Intravenous placebo of 0.9% saline administered over 40 minutes
  Other Names: Placebo
  Arms: Placebo; Sublingual Dexmedetomidine
Drug: Sublingual Placebo — Inert sublingual film
  Other Names: Placebo
  Arms: Intravenous Dexmedetomidine; Placebo

SUMMARY:
This is a pragmatic phase III, randomized, blinded, double placebo-controlled, three-arm trial of elderly patients following cardiac surgery to assess the relationship between nighttime intravenous (IV) and sublingual dexmedetomidine on postoperative delirium and functional outcomes after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Scheduled to undergo a cardiac surgical procedure with cardiopulmonary bypass
* Planned postoperative admission to the intensive care unit (ICU)

Exclusion Criteria:

* Allergy or hypersensitivity to dexmedetomidine or the placebo study medication
* Preexisting diagnosis of Alzheimer's Disease or Related Dementia, severe cognitive impairment or delirium at baseline
* Severe liver failure (Child-Pugh score > 5)
* Severe deficit(s) due to structural or anoxic brain damage
* Undergoing a surgical procedure requiring total circulatory arrest
* SARS-CoV-2 positive or symptomatic (e.g., fever, cough, loss of taste/smell)
* Blind, deaf, or unable to communicate in English
* Patients experiencing circumstances for which long-term follow-up might be difficult (e.g., homelessness, active psychotic disorder, or substance abuse)
* Co-enrollment in other interventional studies that, in the opinion of the site investigator and/or PI, might interfere with study participation, collection, or interpretation of the study data

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Delirium | Postoperative day 1
  The primary outcome will be delirium occurring on postoperative day one. Delirium will be assessed using the Confusion Assessment Method (CAM) twice daily. Delirium will be defined as present if either the morning or afternoon assessment are positive for delirium.

SECONDARY OUTCOMES:
Delirium | Postoperative Day 1 to Day 7
  Postoperative delirium will also be assessed as a secondary outcome assessed within the first three days after surgery, and separately within the first seven days following surgery. Delirium will be assessed using the CAM in the same fashion as the primary outcome. In the event the patient is reintubated the CAM-ICU may also be used to assess for postoperative delirium as a secondary outcome.
Delirium Severity | Postoperative day 1 to day 7
  Delirium severity will be assessed using the CAM-Severity (CAM-S) within the first three days following surgery, and separately within the first seven days following surgery. The CAM-S ranges from 0 (no delirium features) to 19, with higher scores indicating worsening delirium severity.
Telephonic Montreal Cognitive Assessment | 30, 180 and 365 days
  Global cognitive function will be assessed with the T-MoCA in-hospital and at three time points after hospital discharge. Different versions of the T-MOCA will be administered at each time point to minimize learning effects. The T-MoCA ranges from 0 (worst) to 22 (best) points, does not require visual cues or writing, and importantly, can be administered over the phone.
Global Health | 30, 180 and 365 days
  Global health will be assessed at 30, 180 and 365 days using the Patient Reported Outcome Measurement Information System (PROMIS) 29 Profile version 2.1. This assessment results in several subscale scores, each reported as a t-score.
Pain at Rest and Upon Exertion | Postoperative day 1 to day 7
  Pain will be assessed within the first seven days following surgery, using a trajectory of pain scores at rest and upon exertion/deep breathing. Pain scores will be elicited from patients daily using the Pain Numeric Rating Scale.
Opioid and Analgesic Administration | 48 hours postoperatively
  Outcomes for opioid administration will evaluate the (a) frequency and (b) total consumption, defined as morphine equivalents, in the first 24 and 48 hours postoperatively. These will be captured based off medical record review.
Hospital Length of Stay | Postoperatively until discharge, an average of six days
  Hospital length of stay will be defined as the number of days after surgery until the time of discharge from the hospital.
Intensive Care Unit Length of Stay | Postoperatively until discharge, an average of 24 hours
  Intensive Care Unit (ICU) length of stay will be calculated as the time from discharge from the initial index ICU stay minus the time of admission into the cardiovascular ICU and will be reported in hours.
Readmission | 30 days postoperatively
  Hospital readmission will be evaluated within the first 30 days postoperatively using the Society for Thoracic Surgery database or via patient report during follow up phone calls.
Inpatient Morbidity | 30 days postoperatively
  Major cardiac events will be evaluated within 30 days postoperatively and include stroke, atrial fibrillation and renal failure. These outcomes will be assessed using the Society for Thoracic Surgery database and medical record review.
Mortality | Postoperatively until discharge, an average of six days, and at 30, 180 and 365 days postoperatively
  All-cause mortality will be assessed in-hospital and at 30, 180 and 365 days postoperatively. Mortality will be assessed using a combination of electronic medical record review, Society for Thoracic Surgery database, and family report during the follow up phone calls.

CONTACTS AND LOCATIONS:
Overall Officials: Oluwaseun Johnson-Akeju, MD, Principal Investigator — Massachusetts General Hospital
Locations (14):
- United States (14):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Iowa Carver College of Medicine, Iowa City, Iowa
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Hospital, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF